CLINICAL TRIAL: NCT02623023
Title: Brimonidine/Timolol Fixed Combination Prophylaxis for Intraocular Pressure Elevation Following Intravitreal Injection of Antivascular Endothelial Growth Factor
Brief Title: Prophylaxis for Anti-VEGF-induced IOP Elevation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated prior to enrollment, lack of support.
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PAVE-001
Record Dates: First submitted 2015-08-06; First posted 2015-12-07 (Estimated); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension | interventions — Brimonidine Tartrate, Timolol Maleate Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combigan group (Experimental): Combigan will be administered twice a day on the day before the intraocular injection and once in the morning of the injection
  Interventions: Drug: Combigan
- Refresh tears (Placebo Comparator): Refresh tears will be administered twice a day on the day before the intraocular injection and once in the morning of the injection
  Interventions: Other: Refresh tears

INTERVENTIONS:
Drug: Combigan — brimonidine/timolol fixed combination (Combigan®, Allergan; Dublin, IRL)
  Other Names: (Combigan®
  Arms: Combigan group
Other: Refresh tears — This is a placebo group. Refresh tears®, Allergan; Dublin, IRL, is a lubricant eye drop that keeps they eye hydrated
  Arms: Refresh tears

SUMMARY:
The purpose of our study is to determine the effect of prophylactic treatment with brimonidine/timolol fixed combination (Combigan®, Allergan; Dublin, IRL) or placebo therapy (Refresh tears®, Allergan; Dublin, IRL) on long-term IOP measurements in patients receiving serial intravitreal injection of 0.5 mg ranibizumab (0.05 mL) with six months follow-up. Intraocular pressure measurements will be correlated with changes on ancillary testing (Humphrey 24-2 visual field testing and optical coherence tomography (OCT) of the optic nerve head (ONH). Our study would be the first large, prospective, randomized double-blind placebo-controlled trial to examine the relationship between anti-vascular endothelial growth factor (VEGF) therapy and sustained ocular hypertension.

DETAILED DESCRIPTION:
The recent introduction of antivascular endothelial growth factor (anti-VEGF) agents has quickly progressed to become the standard of care for several ocular diseases. Between 2006 and 2010, anti-VEGF treatment for neovascular age-related macular degeneration (AMD) was initiated in over 620 000 eyes of Medicare beneficiaries in the United States. This paradigm shift in retinal therapy stems from evidence that VEGF regulates angiogenesis and vascular permeability, processes which characterize the pathophysiology of diabetic retinopathy and AMD. Several large multicenter, randomized clinical trials have demonstrated that patients with neovascular AMD and clinically significant macular edema (CSME) benefit from frequent intravitreal anti-VEGF injections, particularly with ranibizumab . Ranibizumab is a humanized monoclonal antibody Fab fragment (IgG1) that inhibits all identified VEGF isoforms, including VEGF165, VEGF121 and VEGF110.

Rigorous study has consistently demonstrated a good relative safety profile for anti-VEGF agents. While transient rise in intraocular pressure (IOP) is a known effect immediately following intravitreal injection (IVI), sustained IOP elevation was not initially reported in patients undergoing anti-VEGF therapy. It was not until post-hoc analysis of the MARINA , ANCHOR AND VIEW trials that a significant long-term effect on IOP from ranibizumab was detected. However, there are increasing reports in the literature documenting this phenomenon.

Bakri et al. reported a case series of ocular hypertension (OHT) (IOP ranging 30 - 50 mm Hg) after 0.05 mL intravitreal ranibizumab, which persisted and required treatment. Kahook et al. published a case series of six patients undergoing anti-VEGF therapy who developed persistent OHT, two of whom had a prior diagnosis of glaucoma/glaucoma suspect. In a larger, retrospective review of 215 patients being treated with IVI by Good et al., 6% of patients required medical or laser treatment for sustained IOP elevation. Subgroup analysis revealed that patients with a history of glaucoma had a substantially higher likelihood of experiencing sustained IOP elevation, despite a lower median number of IVI than the non-glaucoma group. In a retrospective study by Choi et al. , seven of 127 patients (5.5%) developed sustained OHT in the study eye, whereas the fellow eye demonstrated stable IOP. Two other large retrospective series have reported similar incidence of persistent IOP elevation, and review of the literature reveals an incidence of 3.45% to 11.6% in patients with neovascular AMD. Post-hoc analysis of a large, multi-center randomized clinical trial for treatment of diabetic CSME found the ranibizumab group had a 3-fold increased risk of sustained IOP elevation at 3 years compared to the sham-injection group. This study did not enroll patients with a history of glaucoma/glaucoma suspect, thus could not define their risk ratio. A prospective study of 217 eyes undergoing anti-VEGF IVI found that persistent IOP elevation was a frequent outcome, and that the IOP peak was significantly correlated with the number of injections. Further, patients with prior diagnosis of glaucoma/glaucoma suspect had an incidence of 12.9% of sustained OHT, compared with 3.2% in the non-glaucoma subgroup.

The pathogenesis of persistent ocular hypertension has not yet been elucidated, but may be secondary to chemical damage to the trabecular meshwork from the anti-VEGF agents themselves, or mechanically by micro-particle obstruction. Some studies indicate that the number of IVI is an independent risk factor for the development of long-term ocular hypertension , and that patients with pre-existing glaucoma are particularly vulnerable.

Transient IOP elevation following anti-VEGF injection has been noted at 30 minutes post-injection and rarely requires anterior chamber paracentesis for treatment . Though this rise in IOP elevation is expected to return to baseline by 1-hour post-IVI, the long-term consequences of this phenomenon are unknown. One proposed mechanism for this transient effect on IOP is increased volume of intraocular contents after injection . Gismondi et al found a significant relationship between shorter axial length and higher transient IOP following intravitreal ranibizumab. One group designed a randomized controlled trial to evaluate the effect of preventative treatment for this short-term rise in IOP. Brimonidine/timolol fixed combination (Combigan®, Allergan; Dublin, IRL) was administered twice a day on the day prior to injection and on the day of treatment, and reduced the rapid increase in post-injection IOP in a safe and effective manner. However, this study did not evaluate the incidence of persistent OHT.

As IOP elevation is strongly linked with the development of glaucoma, this potential outcome in patients undergoing anti-VEGF therapy warrants attention. The data published on this topic to date is primarily comprised of retrospective chart reviews, case series, and post-hoc analysis of the MARINA, ANCHOR and Diabetic Retinopathy Clinical Research Network 2010 and VIEW trials. Many studies reveal inconsistent methodology in terms of IOP measurement and IVI technique. Ultimately, there is no consensus on which factors may predispose patients to the development of iatrogenic IOP elevation following anti-VEGF therapy. Further, prophylactic treatment for sustained OHT has not been prospectively studied.

Currently, there are no guidelines for IOP monitoring in patients undergoing anti-VEGF therapy. Our study aims to define a treatment algorithm for the monitoring and prophylaxis of anti-VEGF-related iatrogenic ocular hypertension. This may also shed some light into the possible mechanism of post-injection IOP spike. Further, our research may help identify a subgroup of patients vulnerable to long-term sequelae as a result of this phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* Baseline visual acuity between 20/40 and 20/200 in the eye chart score
* Diagnosed with either, CNV secondary to neovascular AMD, CSME secondary to diabetes mellitus (DM), or CSME secondary to retinal vein occlusion (RVO)

Exclusion Criteria:

* Baseline IOP ≥30 mmHg
* Diagnosed with Neovascular glaucoma
* Patients unable to undergo Humphrey 24-2 visual field testing or optical coherence tomography
* Active ocular inflammatory disease including uveitis
* Prior retinal or vitreous surgery including vitrectomy, gas tamponade, silicone oil tamponade or scleral buckling
* Prior surgical management of glaucoma including trabeculectomy or filtering device
* Active hepatitis or clinically significant liver disease
* Clinically significant kidney disease
* History of penetrating injury or severe ocular trauma
* Concurrent enrolment in other clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
long-term intraocular pressure measurements | 6 months
  long-term IOP measurements in patients receiving serial IVI of 0.5 mg ranibizumab (0.05 mL) with six months follow-up